CLINICAL TRIAL: NCT02997579
Title: Prospective Randomized Controlled Trial: Comparison of Vibration Arthrometry Between Patella Resurfacing and Patella Non-resurfacing in Total Knee Replacement Patients
Brief Title: Comparison of Vibration Arthrometry Between Patella Resurfacing and Patella Non-resurfacing in Total Knee Replacement Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Satit Thiengwittayaporn, Associate Professor, Navamindradhiraj University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: COA113/2559
Record Dates: First submitted 2016-12-10; First posted 2016-12-20 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Patellar Crepitus; Vibroacoustic Signal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patellar resurfacing (Experimental): patellar resurfacing TKA
  Interventions: Procedure: patellar resurfacing
- patellar non-resurfacing (No Intervention): patellar non-resurfacing TKA

INTERVENTIONS:
Procedure: patellar resurfacing — patellar component insert with cement
  Arms: patellar resurfacing

SUMMARY:
Patellar crepitus is a complication of total knee arthroplasty (TKA).The development of patellar crepitus after TKA are related to many factors such as femoral component design, surgical errors, and postoperative patellar baja. However, it is unclear whether patella resurfacing or patella non-resurfacing are associate with patellar crepitus. The primary objective of this study are to compare the prevalence of patellar crepitus and the mean value of vibroacoustic signal between patellar-resurfacing and patellar non-resurfacing in TKA. The secondary objective is to study the association between patellar crepitus and vibroacoustic signal.

ELIGIBILITY:
Inclusion Criteria:

* primary osteoarthritis of knee

Exclusion Criteria:

* rheumatoid arthritis
* morbid obesity
* severe patellofemoral joint destruction
* patella maltracking
* patellofemoral incongruent
* inflammatory arthritis
* refuse to participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
change of patellar crepitus | pre-op, 3, 6 month
  patellar crepitus investigate by physical examination
change of mean of vibroacoustic signal | pre-op, 3, 6 month

SECONDARY OUTCOMES:
Number of patellar crepitus related to mean of vibroacoustic signal | pre-op, 3, 6 month
  study the association between patellar crepitus and vibroacoustic signal, patellar crepitus investigate by physical examination and mean of vibroacoustic signal assessed by an acceleration sensor

CONTACTS AND LOCATIONS:
Overall Officials: Satit Thiengwittayaporn, M.D., Principal Investigator — Department of Orthopaedics, Faculty of Medicine Vajira Hospital, Navamindradhiraj University
Locations (1):
- Navamindradhiraj University, Dusit, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baczkowicz D, Majorczyk E. Joint motion quality in vibroacoustic signal analysis for patients with patellofemoral joint disorders. BMC Musculoskelet Disord. 2014 Dec 12;15:426. doi: 10.1186/1471-2474-15-426. PMID 25496721
- [Background] Tanaka N, Hoshiyama M. Vibroarthrography in patients with knee arthropathy. J Back Musculoskelet Rehabil. 2012;25(2):117-22. doi: 10.3233/BMR-2012-0319. PMID 22684203